CLINICAL TRIAL: NCT00837746
Title: Bone Histomorphometry, Microarchitecture, and Matrix Structure in Patients Receiving Risedronate Daily or Weekly
Brief Title: Analysis of Iliac Crest Biopsies From Patients Receiving Risedronate
Status: Completed | Type: Observational
Sponsor: Warner Chilcott (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: 2004140
Record Dates: First submitted 2009-02-03; First posted 2009-02-05 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Risedronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Women taking risedronate for 5 years
  Interventions: Drug: risedronate

INTERVENTIONS:
Drug: risedronate — risedronate tablet, 5 mg daily or 35 mg once weekly for 5 years

SUMMARY:
This study analysed and reported on the study data from three similar, risedronate studies, 1996052, 2003073, and 2003096. The objective of the study was to determine the differences in the iliac crest bone histomorphometry and bone quality in postmenopausal women who had received long term therapy with risedronate.

ELIGIBILITY:
Inclusion Criteria:

* Completed month 36 of Study RVN-008993.
* Underwent an iliac crest bone biopsy at month 36.

Exclusion Criteria:

* Was less than 60% compliant with regard to taking study drug from the start of the study drug to month 24 of study RVN-008993.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2003-04; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Differences in iliac crest bone histomorphometry and bone quality in patients receiving risedronate | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Ana M Balske, MD, Study Director — Procter and Gamble
Locations (8):
- United States (7):
  - Maria Greenwald, MD, Palm Desert, California
  - Paul Miller, MD, Lakewood, Colorado
  - Grattan Woodson, MD, Decatur, Georgia
  - Christopher Recknor, MD, Gainesville, Georgia
  - Robert Recker, MD, Omaha, Nebraska
  - Nelson Watts, MD, Cincinnati, Ohio
  - Ronald D Emkey, MD, Wyomissing, Pennsylvania
- Louis-Georges Ste-Marie, MD, Montreal, Quebec, Canada